CLINICAL TRIAL: NCT05635825
Title: Energy and Nutrient Profiles When Asians Transit From a Meat-based to a Plant-based Diet: A Modelling Exercise
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Prince September Pte Ltd Singapore (Unknown)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Other Study IDs: 2021-110
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Nutrition, Healthy
Keywords: plant-based alternative protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Asian: Healthy Asian, non-vegetarian that is aged between 21 to 99, literate and numerate.
  Interventions: Other: Observational Survey

INTERVENTIONS:
Other: Observational Survey — Collection of a 4-day food record

SUMMARY:
This study aims to model and present a simulation exercise to assess the nutritional effects of replacing meat-based protein with meat analogues. The hypothesis of our study is to understand if any positive or detrimental effects on nutrition and health will ensue, when people replace a meat-based diet with plant-based and alternative protein substitutes.

DETAILED DESCRIPTION:
A total of up 100 participants (Chinese/Malay/Indian), non-vegetarians, aged between 21 to 99 years, literate and numerate will be recruited for this study. Participants will be required to complete a 4-day food record as part of the exercise. To ensure accuracy of food records, participants will be requested to either weigh their foods or take photographs of all food and drink consumed during the duration of the study. After all the food records have been collected, the data will be analysed using food composition tables. Nutritional profiles of all participants will be generated. Animal-based products will then be substituted with plant-based counterparts and a new nutritional profile will be generated for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* 21-99 years old
* Non-vegetarians
* Access to smart phone devices if participants intend to use photographic methods

Exclusion Criteria:

* Non-english speaking
* Members of any vulnerable populations
* Members of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted

Ages: 21 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy Asian, non-vegetarian, literate and numerate participants aged between 21-99 years.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Protein | 4 days
  Food record of dietary protein intake
Carbohydrates | 4 days
  Food record of carbohydrate intake
Fats | 4 days
  Food record of fat intake
Minerals | 4 days
  Food record of mineral intake
Dietary fibre | 4 days
  Food record of dietary fibre intake
Cholesterol | 4 days
  Food record of cholesterol intake

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No